CLINICAL TRIAL: NCT00856024
Title: ATHENAS - Retrospective Analysis of Compliance to Treatment of Chronic Hepatitis C With Pegylated Interferon Alpha 2b Associated to Ribavirin Until Week 12 and Correlation With Virological Response in Brazil Health Centers
Brief Title: ATHENAS - Retrospective Study of Compliance in Chronic Hepatitis C With Pegylated Interferon Alfa-2b/Ribavirin in Brazil (P05632)
Acronym: ATHENAS
Status: Terminated | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05632; BR 002-07
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Naïve patients: Patients, from Brazil, with confirmed chronic hepatitis C and who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin and who previous to this treatment had not been treated with peginterferon alfa-2b.
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin
- Group 2: Re-treatment: Patients, from Brazil, with confirmed chronic hepatitis C and who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin and who previous to this treatment had been considered nonresponders or relapsing to prior treatment for chronic hepatitis C.
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin
- Group 3: HIV/HCV co-infected patients: Patients, from Brazil, with confirmed chronic hepatitis C and infected with Humman Immunodeficiency Virus (HIV) who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin.
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alfa-2b — PegIntron 80 μg, PegIntron 100 μg, or PegIntron 120 μg. The duration of the complete treatment and the doses of pegylated interferon alfa 2b should have been prescribed according to local guidelines, and according to the investigating physician's orientation.
  Other Names: SCH 54031
Drug: Ribavirin — Ribavirin 250 mg. The duration of the complete treatment and the doses of ribavirin should have been prescribed according to local guidelines, and according to the investigating physician's orientation.
  Other Names: SCH 18908

SUMMARY:
This is a Phase 4, retrospective and observational, multicenter, national (Brazil), open, noncomparative, and nonrandomized study, which does not have visits. This study will be conducted in accordance to Good Clinical Practices. The procedure will be the review of medical records of patients who have already completed 12 weeks of treatment of chronic hepatitis C with peginterferon alfa-2b and ribavirin. This review will take place after the subjects have signed the informed consent form authorizing collection of these data. The collection of data for virological response after Week 12 will be collected prospectively through the review of medical records after the subjects have completed their entire treatment and follow-up period.

DETAILED DESCRIPTION:
This is a Phase 4, retrospective and observational, multicenter, national (Brazil), open, noncomparative, and nonrandomized study, which does not have visits. This study will be conducted in accordance to Good Clinical Practices. The procedure will be the review of medical records of patients who have already completed 12 weeks of treatment of chronic hepatitis C with peginterferon alfa-2b and ribavirin. This review will take place after the subjects have signed the informed consent form authorizing collection of these data. The physician will be filling out the case report form with the information contained in the medical record. Any dose reduction and/or doses not taken during this period will be reported through the case report form. The collection of data for virological response after Week 12 (such as virological response at the end of treatment and sustained virological response after follow-up period) will be collected prospectively through the review of medical records after the subjects have completed their entire treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed his/her willingness in participating in this study, after having been informed of all aspects that are pertinent to his/her decision to participate, by signing and dating the informed consent form (ICF) approved by the Institutional Review Board / Independent Ethics Committee on Research (IRB/IEC).
* Adult patients who are 18 years old or above.
* Must have diagnosis of chronic hepatitis C confirmed through positive qualitative or quantitative PCR (polymerase chain reaction) performed prior to initiation of the patient's treatment. This result shall be documented in the patient's records.
* Must have completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin.
* Patients who started treatment for chronic hepatitis C from the year 2008 or later.

Exclusion Criteria:

* Does not confirm his/her willing in participating in this study or refuses to sign the informed consent form.
* Did not start the treatment with peginterferon alfa-2b and ribavirin.
* Patients who have less than 12 weeks of treatment with peginterferon alfa-2b and ribavirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed chronic hepatitis C and who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin. Patients will come from approximately 65 Brazilian sites and should satisfy all inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 902 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- General Peginterferon + Ribavarin: Participants received peginterferon alfa-2b and ribavirin according to local labeling guidelines and according to the investigating physician's orientation.
Period: Overall Study
Arm/Group | General Peginterferon + Ribavarin
Started | 902
Completed | 902
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | General Peginterferon + Ribavarin
Number analyzed (Participants) | 902
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data were only available for 900 participants
  years | 49.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367
  Male | 535
Region of Enrollment [Number; unit: participants]
  Brazil | 902

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Were Compliant to Treatment in the First 12 Weeks
Description: The participant was considered compliant if he/she had administered 80% of the doses of pegylated interferon alpha 2b and 80% of the doses of ribavirin that were prescribed by the physician in the first 12 weeks of treatment.
Time Frame: First 12 weeks of treatment
Population: All enrolled participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Naïve Participants: Participants, from Brazil, with confirmed chronic hepatitis C and who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin and who previous to this treatment had not been treated with peginterferon alfa-2b. Participants received peginterferon alfa-2b and ribavirin according to local labeling guidelines and according to the investigating physician's orientation.
- Re-treatment: Participants, from Brazil, with confirmed chronic hepatitis C and who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin and who previous to this treatment had been considered nonresponders or relapsing to prior treatment for chronic hepatitis C. Participants received peginterferon alfa-2b and ribavirin according to local labeling guidelines and according to the investigating physician's orientation.
- HIV/Hepatitis C Virus (HCV) Co-infected Participants: Participants, from Brazil, with confirmed chronic hepatitis C and infected with human immunodeficiency virus (HIV) who completed 12 weeks of treatment with peginterferon alfa-2b and ribavirin. Participants received peginterferon alfa-2b and ribavirin according to local labeling guidelines and according to the investigating physician's orientation.
Arm/Group | Naïve Participants | Re-treatment | HIV/Hepatitis C Virus (HCV) Co-infected Participants
Number analyzed (Participants) | 669 | 199 | 34
Percent of participants | 98.5 [97.3 to 99.3] | 98.5 [95.7 to 99.7] | 100.0 [89.7 to 100.0]

2. Secondary Outcome: Percent of Participants Who Achieved Rapid Virologic Response (RVR)
Description: RVR was defined as HCV RNA negative after 4 weeks of treatment.
Time Frame: Week 4
Population: Number of participants with data
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Naïve Participants | Re-treatment | HIV/Hepatitis C Virus (HCV) Co-infected Participants
Number analyzed (Participants) | 170 | 48 | 6
Percent of participants | 34.7 [27.6 to 42.4] | 18.8 [8.9 to 32.6] | 0.0 [0.0 to 45.9]

3. Secondary Outcome: Percent of Participants Who Achieved Early Virologic Response (EVR)
Description: EVR was defined as HCV RNA negative after 12 weeks of treatment.
Time Frame: Week 12
Population: Number of participants with data
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Naïve Participants | Re-treatment | HIV/Hepatitis C Virus (HCV) Co-infected Participants
Number analyzed (Participants) | 118 | 32 | 6
Percent of participants | 67.8 [58.6 to 76.1] | 46.9 [29.1 to 65.3] | 33.3 [4.3 to 77.7]

ADVERSE EVENTS:
Arm/Group | General Peginterferon + Ribavarin
Serious Adverse Events (participants affected / at risk) | 11/902
Other Adverse Events (participants affected / at risk) | 658/902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Peginterferon + Ribavarin (N=902)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General Peginterferon + Ribavarin (N=902)
ANAEMIA (Blood and lymphatic system disorders) | 204 (205)
NEUTROPENIA (Blood and lymphatic system disorders) | 47 (48)
NAUSEA (Gastrointestinal disorders) | 140 (141)
ASTHENIA (General disorders) | 180 (183)
FATIGUE (General disorders) | 123 (124)
INFLUENZA LIKE ILLNESS (General disorders) | 116 (117)
IRRITABILITY (General disorders) | 52 (53)
PYREXIA (General disorders) | 251 (253)
DECREASED APPETITE (Metabolism and nutrition disorders) | 100 (101)
MYALGIA (Musculoskeletal and connective tissue disorders) | 129 (132)
HEADACHE (Nervous system disorders) | 183 (186)
INSOMNIA (Psychiatric disorders) | 54 (54)
PRURITUS (Skin and subcutaneous tissue disorders) | 62 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The text of the article that will be submitted to the journal shall be defined in common accord between the Investigators and the Sponsor. The principal investigators also agree to not publish and/or present interim results of the study without due written authorization of the Sponsor.